CLINICAL TRIAL: NCT00290576
Title: Digestive and Nutritional Effects of Probiotics (Bifidobacterium Longum and Lactobacillus GG) Supplementation in Premature Newborns
Brief Title: Digestive and Nutritional Effects of Probiotics Supplementation in Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BRD/04/2-Y
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Duration of Parenteral Nutrition
Keywords: Digestive and Nutritional Effects; Safety and Growth; Feeding Tolerance

INTERVENTIONS:
Dietary Supplement: Probiotics supplementation until weight reaches 1800g (Bifidobacterium Longum and Lactobacillus GG )

SUMMARY:
Symbiotic interaction between probiotics ("Living alimentary microbials supplemental, affecting positively host by improving intestinal microbial equilibrium" (Fuller, 1989)) and human digestive tract was amply experimented and seems to be an interesting solution to orientate neonates digestive flora. Many studies showed a probant efficiency of probiotic supplementation in neonates on ECUN, despite abnormally high ECUN incidence in control group. Nevertheless, our aim is to test clinical efficiency of two new probiotics strains. Bifidobacterium Longum and Lactobacillus GG on Oral Nutrition (volume at Day 14 and Day 21) and safety (Adverse Events) in very premature babies.

ELIGIBILITY:
Inclusion Criteria:

1. newborns (< 2 weeks of life)
2. 32 Weeks of Gestation,
3. weight < 1500g,
4. Enteral nutrition begun,
5. Clinical stability,
6. Signed consent form from both parents.

Exclusion Criteria:

1. newborns (>= 2 weeks of life),
2. weight >= 1500g,
3. pathology avoiding the start of the enteral nutrition,
4. other pathologies of those due to premature and its complications,
5. No signed consent form.

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Success if Patient reaches 50% of Nutritional needs by Enteral Nutrition | at D14 and D21.

SECONDARY OUTCOMES:
Age when Enteral Nutrition reaches 50% of Nutritional needs.
Incidence of Nosocomial Infections.
Composition of Colic Flora.
Fecal Calprotectin as Index of Inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Bourdon A, Rouge C, Legrand A, Des Robert C, Piloquet H, Vodovar M, Voyer M, Roze JC, Darmaun D. Urinary citrulline in very low birth weight preterm infants receiving intravenous nutrition. Br J Nutr. 2012 Oct;108(7):1150-4. doi: 10.1017/S0007114511006660. Epub 2011 Dec 12. PMID 22152114
- [Derived] Rouge C, Piloquet H, Butel MJ, Berger B, Rochat F, Ferraris L, Des Robert C, Legrand A, de la Cochetiere MF, N'Guyen JM, Vodovar M, Voyer M, Darmaun D, Roze JC. Oral supplementation with probiotics in very-low-birth-weight preterm infants: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2009 Jun;89(6):1828-35. doi: 10.3945/ajcn.2008.26919. Epub 2009 Apr 15. PMID 19369375